CLINICAL TRIAL: NCT00896688
Title: Ultrasound Guided Diagnostic Cervical Medial Branch Block
Status: Withdrawn | Type: Observational
Why Stopped: The PI has been unable to continue with the study.
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: McMaster University (Other)
Responsible Party: Sponsor
Organization: McMaster University (Other)
Other Study IDs: 08-575-D
Record Dates: First submitted 2009-04-30; First posted 2009-05-12 (Estimated); Last update posted 2018-12-14 (Actual); Status verified 2018-12

CONDITIONS: Facet Joint Pain; Neck Pain
Keywords: cervical branch block; fluoroscopic guidance; ultrasound guidance
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy Volunteers: It will involve 5 volunteers and they will undergo C arm fluoroscopic guided cervical medial branch blocks (C2-C7) on unilateral position and then followed by the 3D ultrasound machine for visualization of needle position.
  Interventions: Procedure: cervical medial branch blocks using the Quincke spinal needle
- Candidates for upper and lower cervial medical branch blocks: This will involve 25 patients and they will follow the same procedures as the healthy volunteers.
  Interventions: Procedure: cervical medial branch blocks using the Quincke spinal needle

INTERVENTIONS:
Procedure: cervical medial branch blocks using the Quincke spinal needle — #25 gauge 1 and 1/2 inch long needle and #25 gauge 10cm long Quincke spinal needle will be used for placement.

SUMMARY:
The diagnostic cervical branch block for neck pain due to cervical facet joint pain has been traditionally done under fluoroscopic guidance. Its diagnostic value and technique have been well established. However, recently some studies have shown that the diagnostic cervical and lumbar medial branch block can be done under ultrasound guidance.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers
* patients who have headache, neck pain, and shoulder pain due to possible facet joint disease

Exclusion Criteria:

* patients/volunteers with BMI > 35
* patients/volunteers with short thick neck
* coagulopathy
* allergy to local anesthetic, ultrasound gel
* patient unable to fill out post procedure pain diary

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
To determine the efficacy of the use of ultrasound for diagnostic cervical medial branch block on pain patients who have developed neck pain, cervicogenic headache, or shoulder pain. | At time of procedure

SECONDARY OUTCOMES:
Interventional pain procedure studies on chronic pain patients | At time of procedure

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Park, MD, Principal Investigator — Hamilton Health Sciences Corporation
Locations (1):
- Hamilton Health Sciences, Hamilton, Ontario, Canada

REFERENCES:
- [Background] Fishman SM, Smith H, Meleger A, Seibert JA. Radiation safety in pain medicine. Reg Anesth Pain Med. 2002 May-Jun;27(3):296-305. doi: 10.1053/rapm.2002.32578. No abstract available. PMID 12016604
- [Background] Greher M, Scharbert G, Kamolz LP, Beck H, Gustorff B, Kirchmair L, Kapral S. Ultrasound-guided lumbar facet nerve block: a sonoanatomic study of a new methodologic approach. Anesthesiology. 2004 May;100(5):1242-8. doi: 10.1097/00000542-200405000-00028. PMID 15114223